CLINICAL TRIAL: NCT06211166
Title: Predicting Patient Relapse After Allogeneic Hematopoietic Stem Cell Transplantation: A Comparison of Measurable Residual Disease (MRD) Assessment by Digital Polymerase Chain Reaction and Conventional MRD
Brief Title: Assessment of Measurable Residual Disease in Allo-HSCT Using Digital Polymerase Chain Reaction
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Professor, Peking University People's Hospital
Other Study IDs: 2021PHA154-001
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Acute Leukemia; MDS; MDS/MPN; CML
Keywords: dPCR; MRD; allo-HSCT; leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute Leukemia: Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, Mixed Phenotype Acute Leukemia
  Interventions: Diagnostic Test: Digital PCR; Diagnostic Test: Quantitative PCR; Diagnostic Test: MFC
- MDS or MDS/MPN: Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia, and other subtypes of Myelodysplastic/Myeloproliferative Neoplasm
  Interventions: Diagnostic Test: Digital PCR; Diagnostic Test: Quantitative PCR; Diagnostic Test: MFC
- CML: Chronic Myeloid Leukemia
  Interventions: Diagnostic Test: Digital PCR; Diagnostic Test: Quantitative PCR

INTERVENTIONS:
Diagnostic Test: Digital PCR — digital Polymerase Chain Reaction (dPCR)
Diagnostic Test: Quantitative PCR — Real-time Polymerase Chain Reaction (real-time PCR)
Diagnostic Test: MFC — Multicolor Flow Cytometry
  Groups: Acute Leukemia; MDS or MDS/MPN

SUMMARY:
A research investigation into the efficacy of digital Polymerase Chain Reaction (dPCR) for monitoring measurable residual disease (MRD) during allogeneic hematopoietic stem cell transplantation, with a focus on predicting relapse in patients diagnosed with leukemia, myelodysplastic syndromes (MDS), and related hematological conditions.

DETAILED DESCRIPTION:
This prospective clinical study focuses on patients diagnosed with leukemia, myelodysplastic syndromes (MDS), and related hematological conditions post-allogeneic hematopoietic stem cell transplantation. The primary objective is to assess the efficacy of digital Polymerase Chain Reaction (dPCR) in monitoring measurable residual disease (MRD), including markers such as BCR::ABL, KMT2A, etc., as compared to other MRD monitoring methods such as conventional quantitative PCR or multicolor Flow Cytometry (MFC). Key endpoints include the recurrence of MRD using conventional methods, hematological relapse, disease-free survival, overall survival, and non-relapse mortality.

ELIGIBILITY:
Inclusion Criteria:

* The presence of at least one fusion gene or hematological tumor-associated mutation detected at diagnosis by NGS or real-time PCR provided for posttransplant MRD monitoring.
* Neutrophil engraftment
* Received at least one MRD monitoring by digital PCR after HSCT

Exclusion Criteria:

* Patients who relapsed or died before the first digital PCR monitoring
* Patients only with mutations in DNMT3A, TET2, and ASXL1 ("DTA mutations") or only germline mutations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematological malignancies who underwent allo-HSCT were enrolled for MRD monitoring peri-HSCT
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Threshold of dPCR to predict conventional MRD | 2-year
  To establish an optimal threshold for digital PolyTo establish an optimal threshold for digital Polymerase Chain Reaction (dPCR) in predicting Measurable Residual Disease (MRD) recurrence after allogeneic hematopoietic stem cell transplantation (allo-HSCT). MRD recurrence is defined as the reappearance or elevation of minimal residual disease, as assessed by other MRD monitoring methods such as conventional quantitative PCR or multi-color Flow Cytometry (MFC), which served as indications of pre-emptive intervention by current consensus or guideline.

SECONDARY OUTCOMES:
Cumulative incidence of relapse (CIR) | 2-year
  The interval from the transplantation date to hematological recurrence
Overall survival (OS) | 2-year
  The time from HSCT to the Death from any cause
Relapse-free survival (RFS) | 2-year
  The time from the date of HSCT to the occurrence of any of the following: Death from any cause Disease recurrence
Non-Relapse Mortality(NRM) | 2-year
  The time from the date of HSCT to deaths that result from complications other than a relapse of the underlying disease.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-jun Huang, M.D, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No